CLINICAL TRIAL: NCT05232578
Title: Early Salvage Therapy for Patients With Advanced Features for Biochemical Relapse After Radical Prostatectomy for Localized Prostate Carcinoma In Correlation With Supposed Molecular-genetic Parameters of Higher Aggressiveness
Acronym: ESTABLISH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Sona Argalacsova, Principal Investigator, Radiation oncology head, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESTABLISH 2021 Trial v03.2021
Record Dates: First submitted 2021-11-24; First posted 2022-02-10 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: prostate carcinoma; salvage therapy; biochemical relapse
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A "balanced design" is used for the 1:1 randomization into two arms A and B:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A- early salvage radiotherapy (eSRT) (Experimental): Early salvage radiotherapy (eSRT) will be administered immediately after the confirmation of the biochemical relapse (prostate-specific antigen PSA level increase to ≈ 0,2 ng/ml) after radical prostatectomy with defined risk factors and no clinical recurrence signs on prostate specific membrane antigen positron emission tomography and computed tomography (PSMA PET/CT).
  Interventions: Radiation: Early salvage radiotherapy (eSRT)
- Arm B- delayed salvage radiotherapy (dSRT) (Experimental): The patient is by the biochemical relapse analysis (PSA level 0,2 ng/ml) referred for further follow-up of PSA values. dSRT is initiated, if PSA further increase to values of ≥ 0.4 ng/ml is confirmed and the presence of a potential clinical relapse is excluded with repeated PSMA-PET-CT in line with standard procedures
  Interventions: Radiation: Delayed Salvage radiotherapy (dSRT)

INTERVENTIONS:
Radiation: Early salvage radiotherapy (eSRT) — eSRT administered immediately after the confirmation of the biochemical relapse (PSA ≈ 0.2ng/ml).
  66-70Gy will be delivered to the bed of prostate. Radiotherapy will be optionally accompanied by androgen deprivation therapy.
  Arms: Arm A- early salvage radiotherapy (eSRT)
Radiation: Delayed Salvage radiotherapy (dSRT) — dSRT administered if PSA levels increase to ≥ 0.4 ng/ml.
  66-70Gy will be delivered to the bed of prostate. Radiotherapy will be optionally accompanied by androgen deprivation therapy.
  Arms: Arm B- delayed salvage radiotherapy (dSRT)

SUMMARY:
The primary objective of the trial is to compare the impact and safety of delayed salvage therapy (dSRT, i.e., SRT initiated at PSA values of 0.4-0.5 ng/ml) to those of early salvage therapy (eSRT, i.e., at PSA levels of 0.2 ng/ml) in patients with biochemical relapse after radical prostatectomy.

The secondary objective of the trial is to perform analysis of the subgroups of patients to determine which patients are most likely to benefit from dSRT

Exploratory objective of the trial is to determine whether selected molecular genetic parameters (172 candidate genes and molecular alterations) and known clinical parameters can be used to identify potential predictors of worse prognosis in patients with known risk factors for relapse after radical prostatectomy, thereby augmenting and refining patient stratification, optimizing their therapy, and clarifying the proper timing of multimodal therapy

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Pathologically confirmed invasive prostate carcinoma with minimal 1 risk factor (RF) after radical prostatectomy (RP)
* Patient refuses the adjuvant therapy after normalization of urinary function within 6 month after RP
* Signed informed consent to participate in the study and (where necessary) consent to participate in the translational part of the research (not a requirement)
* ECOG 0 - 1
* pT2 and minimal 1 risk factor (RF):

  * R1 (PSM), and/or
  * Gleason score (4+3=7) 8-10 and/or ISUP grade group 3-5
* pT3a /pT3b with or without one RF
* No evidence of suspicious pelvic lymph nodes by initial diagnostic: cN0 and/or pN0
* No evidence of suspicious distant metastases by initial diagnostic: M0
* Patient with decline of PSA level to undetectable PSA levels (< 0,1 ng/ml) or around 0,2ng/ml and with another decreasing trends so that the PSA level decline within 12-24 weeks after RP to undetectable levels (< 0,1 ng/ml) and with renewed increase of PSA >0,2 ng/ml (BCR= biochemical relapse) without any clinical relapse on PSMA PET/CT
* No hormonal therapy prior and /or after the radical prostatectomy
* Patient suitable and fit for subsequent radiotherapy with high likelihood of good compliance to the follow-up

Exclusion Criteria:

* Life expectancy (based on Charlson comorbidity index) < 10 years
* Patient not fit for the therapy
* History of other cancer (other than a radically removed non-melanoma skin carcinoma)
* Previous pelvic irradiation
* Active immunosuppressive medication
* History of hormone therapy prior to randomization
* cN1 and/or pN1 and M1
* PSA-persistence after RP (PSA 12-weeks after RP > 0.1 ng/ml or no decreasing trend described in Inclusion criteria)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Analysed 3 years after randomisation of the last patient.
  Defined as a time to re-documented biochemical relapse after salvage therapy (bRFS), demonstration of clinical relapse (i.e.,local relapse /lRFS/, locoregional relapse /lrRFS/, distant relapse /MFS/) and/or death from any cause.

SECONDARY OUTCOMES:
Carcinoma-specific survival (CSS) | Analysed 5/10 years after randomization of the last patient.
Overall survival (5y- and 10y- OS) | Analysed 5/10 years after randomization of the last patient.
Incidence of treatment-related acute and late toxicity | Analysed 5 years after randomization of the last patient.
  Comparison of the incidence of treatment-related acute and late toxicity between patients after early/ delayed salvage therapy.
  Acute and late toxicity will be assessed and graded using Common Terminology Criteria for Adverse Events (CTCAE).
Health-related quality of life (QoL) assessment. | Analysed 5 years after randomization of the last patient.
  The analysis of the QoL of both study ARMs will be made based on EORTC validated questionnaires (QLQ-C30 and QLQ-PR25).
  QLQ-C30 was developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. The EORTC QLQ-PR25 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 25 items specifically related to prostate cancer.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kneebone A, Fraser-Browne C, Duchesne GM, Fisher R, Frydenberg M, Herschtal A, Williams SG, Brown C, Delprado W, Haworth A, Joseph DJ, Martin JM, Matthews JHL, Millar JL, Sidhom M, Spry N, Tang CI, Turner S, Wiltshire KL, Woo HH, Davis ID, Lim TS, Pearse M. Adjuvant radiotherapy versus early salvage radiotherapy following radical prostatectomy (TROG 08.03/ANZUP RAVES): a randomised, controlled, phase 3, non-inferiority trial. Lancet Oncol. 2020 Oct;21(10):1331-1340. doi: 10.1016/S1470-2045(20)30456-3. PMID 33002437
- [Background] Tao R, Dai J, Bai Y, Yang J, Sun G, Zhang X, Zhao J, Zeng H, Shen P. The prognosis benefits of adjuvant versus salvage radiotherapy for patients after radical prostatectomy with adverse pathological features: a systematic review and meta-analysis. Radiat Oncol. 2019 Nov 9;14(1):197. doi: 10.1186/s13014-019-1384-z. PMID 31706339
- [Background] Wiegel T, Bartkowiak D, Bottke D, Bronner C, Steiner U, Siegmann A, Golz R, Storkel S, Willich N, Semjonow A, Stockle M, Rube C, Rebmann U, Kalble T, Feldmann HJ, Wirth M, Hofmann R, Engenhart-Cabillic R, Hinke A, Hinkelbein W, Miller K. Adjuvant radiotherapy versus wait-and-see after radical prostatectomy: 10-year follow-up of the ARO 96-02/AUO AP 09/95 trial. Eur Urol. 2014 Aug;66(2):243-50. doi: 10.1016/j.eururo.2014.03.011. Epub 2014 Mar 21. PMID 24680359
- [Background] Bhindi B, Lokeshwar SD, Klaassen Z, Klotz L, Wallis CJD. Systematic review and meta-analysis of trials evaluating the role of adjuvant radiation after radical prostatectomy for prostate cancer: Implications for early salvage. Can Urol Assoc J. 2020 Oct;14(10):330-336. doi: 10.5489/cuaj.6440. PMID 32432529
- [Background] Bolla M, van Poppel H, Tombal B, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Colombel M, van de Beek C, Verhagen P, van den Bergh A, Sternberg C, Gasser T, van Tienhoven G, Scalliet P, Haustermans K, Collette L; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Genito-Urinary Groups. Postoperative radiotherapy after radical prostatectomy for high-risk prostate cancer: long-term results of a randomised controlled trial (EORTC trial 22911). Lancet. 2012 Dec 8;380(9858):2018-27. doi: 10.1016/S0140-6736(12)61253-7. Epub 2012 Oct 19. PMID 23084481
- [Background] Hackman G, Taari K, Tammela TL, Matikainen M, Kouri M, Joensuu T, Luukkaala T, Salonen A, Isotalo T, Petas A, Hendolin N, Bostrom PJ, Aaltomaa S, Lehtoranta K, Hellstrom P, Riikonen J, Korpela M, Minn H, Kellokumpu-Lehtinen PL, Pukkala E, Hemminki A; FinnProstate Group. Randomised Trial of Adjuvant Radiotherapy Following Radical Prostatectomy Versus Radical Prostatectomy Alone in Prostate Cancer Patients with Positive Margins or Extracapsular Extension. Eur Urol. 2019 Nov;76(5):586-595. doi: 10.1016/j.eururo.2019.07.001. Epub 2019 Jul 30. PMID 31375279
- [Background] Sanda MG, Cadeddu JA, Kirkby E, Chen RC, Crispino T, Fontanarosa J, Freedland SJ, Greene K, Klotz LH, Makarov DV, Nelson JB, Rodrigues G, Sandler HM, Taplin ME, Treadwell JR. Clinically Localized Prostate Cancer: AUA/ASTRO/SUO Guideline. Part II: Recommended Approaches and Details of Specific Care Options. J Urol. 2018 Apr;199(4):990-997. doi: 10.1016/j.juro.2018.01.002. Epub 2018 Jan 10. PMID 29331546
- [Background] McClelland S 3rd, Sandler KA, Degnin C, Chen Y, Mitin T. Adjuvant vs. salvage radiation therapy in men with high-risk features after radical prostatectomy: Survey of North American genitourinary expert radiation oncologists. Can Urol Assoc J. 2019 May;13(5):E132-E134. doi: 10.5489/cuaj.5470. Epub 2018 Oct 15. PMID 30332590
- [Background] Ploussard G, Staerman F, Pierrevelcin J, Saad R, Beauval JB, Roupret M, Audenet F, Peyromaure M, Delongchamps NB, Vincendeau S, Fardoun T, Rigaud J, Villers A, Bastide C, Soulie M, Salomon L; Committee of Cancerology of the Association of French Urology. Predictive factors of oncologic outcomes in patients who do not achieve undetectable prostate specific antigen after radical prostatectomy. J Urol. 2013 Nov;190(5):1750-6. doi: 10.1016/j.juro.2013.04.073. Epub 2013 Apr 30. PMID 23643600
- [Background] Parker CC, Clarke NW, Cook AD, Kynaston HG, Petersen PM, Catton C, Cross W, Logue J, Parulekar W, Payne H, Persad R, Pickering H, Saad F, Anderson J, Bahl A, Bottomley D, Brasso K, Chahal R, Cooke PW, Eddy B, Gibbs S, Goh C, Gujral S, Heath C, Henderson A, Jaganathan R, Jakobsen H, James ND, Kanaga Sundaram S, Lees K, Lester J, Lindberg H, Money-Kyrle J, Morris S, O'Sullivan J, Ostler P, Owen L, Patel P, Pope A, Popert R, Raman R, Roder MA, Sayers I, Simms M, Wilson J, Zarkar A, Parmar MKB, Sydes MR. Timing of radiotherapy after radical prostatectomy (RADICALS-RT): a randomised, controlled phase 3 trial. Lancet. 2020 Oct 31;396(10260):1413-1421. doi: 10.1016/S0140-6736(20)31553-1. Epub 2020 Sep 28. PMID 33002429
- [Background] Vale CL, Fisher D, Kneebone A, Parker C, Pearse M, Richaud P, Sargos P, Sydes MR, Brawley C, Brihoum M, Brown C, Chabaud S, Cook A, Forcat S, Fraser-Browne C, Latorzeff I, Parmar MKB, Tierney JF; ARTISTIC Meta-analysis Group. Adjuvant or early salvage radiotherapy for the treatment of localised and locally advanced prostate cancer: a prospectively planned systematic review and meta-analysis of aggregate data. Lancet. 2020 Oct 31;396(10260):1422-1431. doi: 10.1016/S0140-6736(20)31952-8. Epub 2020 Sep 28. PMID 33002431
- [Background] Sargos P, Chabaud S, Latorzeff I, Magne N, Benyoucef A, Supiot S, Pasquier D, Abdiche MS, Gilliot O, Graff-Cailleaud P, Silva M, Bergerot P, Baumann P, Belkacemi Y, Azria D, Brihoum M, Soulie M, Richaud P. Adjuvant radiotherapy versus early salvage radiotherapy plus short-term androgen deprivation therapy in men with localised prostate cancer after radical prostatectomy (GETUG-AFU 17): a randomised, phase 3 trial. Lancet Oncol. 2020 Oct;21(10):1341-1352. doi: 10.1016/S1470-2045(20)30454-X. PMID 33002438
- [Background] Shipley WU, Seiferheld W, Lukka HR, Major PP, Heney NM, Grignon DJ, Sartor O, Patel MP, Bahary JP, Zietman AL, Pisansky TM, Zeitzer KL, Lawton CA, Feng FY, Lovett RD, Balogh AG, Souhami L, Rosenthal SA, Kerlin KJ, Dignam JJ, Pugh SL, Sandler HM; NRG Oncology RTOG. Radiation with or without Antiandrogen Therapy in Recurrent Prostate Cancer. N Engl J Med. 2017 Feb 2;376(5):417-428. doi: 10.1056/NEJMoa1607529. PMID 28146658
- [Background] Carrie C, Magne N, Burban-Provost P, Sargos P, Latorzeff I, Lagrange JL, Supiot S, Belkacemi Y, Peiffert D, Allouache N, Dubray BM, Servagi-Vernat S, Suchaud JP, Crehange G, Guerif S, Brihoum M, Barbier N, Graff-Cailleaud P, Ruffion A, Dussart S, Ferlay C, Chabaud S. Short-term androgen deprivation therapy combined with radiotherapy as salvage treatment after radical prostatectomy for prostate cancer (GETUG-AFU 16): a 112-month follow-up of a phase 3, randomised trial. Lancet Oncol. 2019 Dec;20(12):1740-1749. doi: 10.1016/S1470-2045(19)30486-3. Epub 2019 Oct 16. PMID 31629656
- [Background] Fossati N, Robesti D, Karnes RJ, Soligo M, Boorjian SA, Bossi A, Coraggio G, Di Muzio N, Cozzarini C, Noris Chiorda B, Gandaglia G, Scarcella S, Bartkowiak D, Bohmer D, Shariat S, Goldner G, Battaglia A, Joniau S, Haustermans K, De Meerleer G, Fonteyne V, Ost P, Van Poppel H, Montorsi F, Wiegel T, Briganti A. Assessing the Role and Optimal Duration of Hormonal Treatment in Association with Salvage Radiation Therapy After Radical Prostatectomy: Results from a Multi-Institutional Study. Eur Urol. 2019 Oct;76(4):443-449. doi: 10.1016/j.eururo.2019.02.004. Epub 2019 Feb 22. PMID 30799187
- [Background] King CR. The timing of salvage radiotherapy after radical prostatectomy: a systematic review. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):104-11. doi: 10.1016/j.ijrobp.2011.10.069. Epub 2012 Jul 14. PMID 22795730
- [Background] Ohri N, Dicker AP, Trabulsi EJ, Showalter TN. Can early implementation of salvage radiotherapy for prostate cancer improve the therapeutic ratio? A systematic review and regression meta-analysis with radiobiological modelling. Eur J Cancer. 2012 Apr;48(6):837-44. doi: 10.1016/j.ejca.2011.08.013. Epub 2011 Sep 22. PMID 21945099
- [Background] Pfister D, Bolla M, Briganti A, Carroll P, Cozzarini C, Joniau S, van Poppel H, Roach M, Stephenson A, Wiegel T, Zelefsky MJ. Early salvage radiotherapy following radical prostatectomy. Eur Urol. 2014 Jun;65(6):1034-43. doi: 10.1016/j.eururo.2013.08.013. Epub 2013 Aug 15. PMID 23972524
- [Background] Abugharib A, Jackson WC, Tumati V, Dess RT, Lee JY, Zhao SG, Soliman M, Zumsteg ZS, Mehra R, Feng FY, Morgan TM, Desai N, Spratt DE. Very Early Salvage Radiotherapy Improves Distant Metastasis-Free Survival. J Urol. 2017 Mar;197(3 Pt 1):662-668. doi: 10.1016/j.juro.2016.08.106. Epub 2016 Sep 7. PMID 27614333
- [Background] Moreira DM, Presti JC Jr, Aronson WJ, Terris MK, Kane CJ, Amling CL, Freedland SJ. Natural history of persistently elevated prostate specific antigen after radical prostatectomy: results from the SEARCH database. J Urol. 2009 Nov;182(5):2250-5. doi: 10.1016/j.juro.2009.07.022. Epub 2009 Sep 16. PMID 19758614
- [Background] Xiang C, Liu X, Chen S, Wang P. Prediction of Biochemical Recurrence Following Radiotherapy among Patients with Persistent PSA after Radical Prostatectomy: A Single-Center Experience. Urol Int. 2018;101(1):47-55. doi: 10.1159/000488536. Epub 2018 Apr 6. PMID 29627830
- [Background] Van den Broeck T, van den Bergh RCN, Arfi N, Gross T, Moris L, Briers E, Cumberbatch M, De Santis M, Tilki D, Fanti S, Fossati N, Gillessen S, Grummet JP, Henry AM, Lardas M, Liew M, Rouviere O, Pecanka J, Mason MD, Schoots IG, van Der Kwast TH, van Der Poel HG, Wiegel T, Willemse PM, Yuan Y, Lam TB, Cornford P, Mottet N. Prognostic Value of Biochemical Recurrence Following Treatment with Curative Intent for Prostate Cancer: A Systematic Review. Eur Urol. 2019 Jun;75(6):967-987. doi: 10.1016/j.eururo.2018.10.011. Epub 2018 Oct 17. PMID 30342843
- [Background] Pound CR, Partin AW, Eisenberger MA, Chan DW, Pearson JD, Walsh PC. Natural history of progression after PSA elevation following radical prostatectomy. JAMA. 1999 May 5;281(17):1591-7. doi: 10.1001/jama.281.17.1591. PMID 10235151
- [Background] Boorjian SA, Thompson RH, Tollefson MK, Rangel LJ, Bergstralh EJ, Blute ML, Karnes RJ. Long-term risk of clinical progression after biochemical recurrence following radical prostatectomy: the impact of time from surgery to recurrence. Eur Urol. 2011 Jun;59(6):893-9. doi: 10.1016/j.eururo.2011.02.026. Epub 2011 Feb 22. PMID 21388736
- [Background] Kristiansen G. Markers of clinical utility in the differential diagnosis and prognosis of prostate cancer. Mod Pathol. 2018 Jan;31(S1):S143-155. doi: 10.1038/modpathol.2017.168. PMID 29297492
- [Background] Bostrom PJ, Bjartell AS, Catto JW, Eggener SE, Lilja H, Loeb S, Schalken J, Schlomm T, Cooperberg MR. Genomic Predictors of Outcome in Prostate Cancer. Eur Urol. 2015 Dec;68(6):1033-44. doi: 10.1016/j.eururo.2015.04.008. Epub 2015 Apr 23. PMID 25913390
- [Background] Robin S, Jolicoeur M, Palumbo S, Zilli T, Crehange G, De Hertogh O, Derashodian T, Sargos P, Salembier C, Supiot S, Udrescu C, Chapet O. Prostate Bed Delineation Guidelines for Postoperative Radiation Therapy: On Behalf Of The Francophone Group of Urological Radiation Therapy. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1243-1253. doi: 10.1016/j.ijrobp.2020.11.010. Epub 2020 Nov 10. PMID 33186618